CLINICAL TRIAL: NCT04594863
Title: The Investigation of the Mechanism of Cachexia Occurrence for Patients With Gastrointestinal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-2525
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — peripheral blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cachexia: patients suffering from cachexia recently
- no cachexia: patients are not suffering from cachexia recently

SUMMARY:
The study is going to recruit patients with gastrointestinal cancer, collect clinical data and peripheral blood sample and possible fat samples. The expression of SIRT-6 in peripheral blood will be tested and connect with different status of cachexia of the patients. A mathematical model of the relationship between cachexia classification and SIRT-6 expression is going to constructed as anticipated.

DETAILED DESCRIPTION:
At the start of cancer develop, not all patients with gastrointestinal cancer manifest cachexia, it may be associated with SIRT-6 expression. This study will collect and test the peripheral blood sample of patients, use it as an important indicator of the degree of cachexia, and provide references for clinical drug intervention, prognosis and dietary intervention for cachexia patients. If possible, fat sample of the patients will be collected during surgery, and the adipose progenitor cells will be cultured to find the key target proteins by detecting differences in protein expression, changes in protein modification levels, and protein interactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 90 years old, unlimited gender;
2. Patients who are diagnosed with gastrointestinal cancer for the first time and are planning to undergo further treatment;
3. Volunteer to participate and sign the informed consent form.

Exclusion Criteria:

1. Women who are pregnant or lactate;
2. Patients with severe metabolic diseases; combined with cardiac function, liver and kidney dysfunction, acute myocardial infarction and acute stroke in the past 3 months , COPD acute onset respiratory failure and other serious medical diseases and patients who need hormone therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with gastrointestinal cancer for the first time without any chemotherapy or radiotherapy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
SIRT-6 expression | 4 months
  SIRT-6 expression tested by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospita, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Argiles JM, Busquets S, Stemmler B, Lopez-Soriano FJ. Cancer cachexia: understanding the molecular basis. Nat Rev Cancer. 2014 Nov;14(11):754-62. doi: 10.1038/nrc3829. Epub 2014 Oct 9. PMID 25291291
- [Background] Fearon KC, Glass DJ, Guttridge DC. Cancer cachexia: mediators, signaling, and metabolic pathways. Cell Metab. 2012 Aug 8;16(2):153-66. doi: 10.1016/j.cmet.2012.06.011. Epub 2012 Jul 12. PMID 22795476